CLINICAL TRIAL: NCT04437758
Title: Effects of Hydrolyzed Collagen and Vitamin C on Explosive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1704
Record Dates: First submitted 2020-06-12; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Collagen Synthesis; Rate of Force (RFD) Development
Keywords: exercise; performance; athletes
MeSH Terms: conditions — Motor Activity | interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque packets coded by Sponsor's Product Development
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolyzed collagen and Vitamin C powder mix (Experimental): 20 g hydrolyzed collagen + 50 mg vitamin C (ascorbic acid) pre-packed powder diluted in 250 ml (8 oz) of water
  Interventions: Dietary Supplement: Collagen and Vitamin C powder mix nutritional intervention; Other: Maximum power training exercise
- Maltodextrin powder (Placebo Comparator): 20 g maltodextrin pre-packed powder diluted in 250 ml (8 oz) of water
  Interventions: Other: Maltodextrin placebo powder; Other: Maximum power training exercise

INTERVENTIONS:
Dietary Supplement: Collagen and Vitamin C powder mix nutritional intervention — 20 g collagen + 50 mg vitamin C daily, 60 min prior to exercise
  Arms: Hydrolyzed collagen and Vitamin C powder mix
Other: Maltodextrin placebo powder — 20 g maltodextrin placebo daily, 60 min prior to exercise
  Arms: Maltodextrin powder
Other: Maximum power training exercise — Explosive/power-based exercise training program 3 times/week at home consisting of drop jumps, box jumps, weighted jump squats loaded in a progressive manner weekly for 3 weeks. At baseline and at the end of each of the 3 weeks, measures of explosive performance are assessed in the lab (maximal isometric squat, counter-movement jump and squat jump)

SUMMARY:
Determine whether supplementation with a combined dose of 20 g of hydrolyzed collagen and 50 mg vitamin C, along with a power training exercise program, increases rate of force development (RFD) and performance in athletes

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male athletes between 18-30 years of age
2. Currently participating in sport
3. <3 musculoskeletal injuries in the past year
4. No health or dietary restriction that would be affected by the supplementation protocol

Exclusion Criteria:

1. History of more than 3 musculoskeletal injuries within the past 12 months
2. Health, dietary restriction or diet that would be affected by the supplementation protocol
3. Willing to eat similar dietary pattern the day before baseline testing and each exercise testing/intervention day

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Collagen synthesis varies significantly throughout the menstrual cycle in females. This natural variation would confound the study. Provided this work proves successful, we will aim to perform similar studies in females.
Enrollment: 50 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Maximal rate of force development (RFD) of isometric squat (MIS) | % change from baseline to week 1, week 2 and week 3
  Force (N) over time (msec) for the maximum slope of the first 20% of the movement
Counter-movement jump (CMJ) rate of force development (RFD) | % change from baseline to week 1, week 2 and week 3
  CMJ jump performance N/s/kg
Squat jump height rate of force development (RFD) | % change from baseline to week 1, week 2 and week 3
  Squat jump height performance RFD/kg

OTHER OUTCOMES:
Maximum peak force of maximal isometric squat (MIS) | % change from baseline to week 1, week 2 and week 3
  Peak force (N)
Counter-movement jump (CMJ) net eccentric impulse | % change from baseline to week 1, week 2 and week 3
  Jump performance max N/s/kg (Note: Eccentric is the drop down part of the CMJ)
Counter-movement jump (CMJ) net concentric impulse | % change from baseline to week 1, week 2 and week 3
  Jump performance max N/s/kg (Note: Concentric is the movement upwards of the CMJ)
Leg stiffness assessment | % change from baseline to week 1, week 2 and week 3
  Tendon stiffness mean per kg (N/m/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Functional Molecular Biology Laboratory and Human Performance Laboratory, Davis, California, United States